CLINICAL TRIAL: NCT02454049
Title: Influence of Dietary Nitrate on Paralympics 2016 Time Trial Performance in Swiss Elite Paracycling Athletes
Brief Title: Influence of Dietary Nitrate on Time Trial Performance in Swiss Paracycling Athletes
Acronym: nitrate_TT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-04
Record Dates: First submitted 2015-05-19; First posted 2015-05-27 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Exercise Nutritional Physiology
MeSH Terms: interventions — sodium nitrate; Water

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- beetroot juice (Active Comparator): beetroot juice containing 6mmol nitrate, ingested 3hours before the exercise test
  Interventions: Dietary Supplement: beetroot juice
- sodium nitrate (Active Comparator): 6mmol sodium nitrate dissolved in plain water, ingested 3hours before the exercise test
  Interventions: Dietary Supplement: sodium nitrate
- water (Placebo Comparator): 85ml of plain water, ingested 3 hours before the exercise test
  Interventions: Dietary Supplement: water

INTERVENTIONS:
Dietary Supplement: beetroot juice — 6mmol nitrate
  Arms: beetroot juice
Dietary Supplement: sodium nitrate — 6mmol sodium nitrate
  Arms: sodium nitrate
Dietary Supplement: water — plain water
  Arms: water

SUMMARY:
The aim of this study is to investigate wether beetroot juice or sodium nitrate enhances time trial performance in Swiss paracycling athletes compared to the ingestion of a placebo supplement. Furthermore, the effects of beetroot juice and sodium nitrate on performance will be investigated in spinal cord injured and non-injured athletes.

DETAILED DESCRIPTION:
The influence of dietary nitrate on performance will be tested performing a time trial on a handbike. The time trial will be the same as in the Paralympics 2016 in Rio. The subjects perform three trials and receive another supplement for each trial: beetroot juice with 6mmol nitrate, 6mmol sodium nitrate or plain water (placebo supplement). The time to complete the time trial will be the main outcome parameter.

ELIGIBILITY:
Inclusion Criteria:

* healthy paracycling athletes
* healthy, able-bodied, upper-body trained individuals

Exclusion Criteria:

* female
* smoking
* any medication affecting performance
* medical conditions affecting performance

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
time to perform trial | 3 hours after supplement ingestion

SECONDARY OUTCOMES:
oxygen consumption during time trial performance measured by a metabolic cart (Oxycon Pro) in ml/min/kg | 3 hours after supplement ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Perret, PD PhD, Principal Investigator — Swiss Paraplegic Centre
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland